CLINICAL TRIAL: NCT06510283
Title: Efficacy and Safety of Taitacept in Treatment of Refractory or Recurrent Anti-NMDAR/anti-LGI1 Encephalitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREC2024-KY061
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-06

CONDITIONS: Anti-N-Methyl-D-Aspartate Receptor Encephalitis
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Taitacept treatment group (Experimental): Telitacicept will be subcutaneously injected at a dose of 240mg per week, lasting for at least 24 weeks.
  Interventions: Drug: Taitacept

INTERVENTIONS:
Drug: Taitacept — Telitacicept will be subcutaneously injected at a dose of 240mg per week, lasting for at least 24 weeks.
  Other Names: No other Intervention Names

SUMMARY:
The main objective is to explore the efficacy and safety of Telitacicept in the treatment of refractory/recurrent anti-NMDAR and anti-LGI1 encephalitis.

Through this prospective, single-center, open-label clinical trial, we aim to investigate the effectiveness and safety of Telitacicept in refractory/recurrent anti-NMDAR and anti-LGI1 encephalitis by add-on therapy of Telitacicept combined with traditional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥14 years old, male or female;
2. Symptoms of autoimmune encephalitis (AE) ≤ 9 months prior to enrollment;
3. Diagnosed as autoimmune encephalitis, diagnostic criteria as follows:

   1. Rapid onset (<3 months) of at least four of the following six major symptoms:

      * Abnormal (mental) behavior or cognitive dysfunction
      * Speech dysfunction (verbal urgency, hypospeech, mutism)
      * Seizures
      * Movement disorders, dyskinesias, or postural rigidity/abnormalities
      * Decreased level of consciousness
      * Autonomic dysfunction or central hypoventilation in the presence of one or more of the six major symptoms;
   2. Positive anti-NMDAR (GluN1) IgG antibody detected in CSF or positive serum and/or cerebrospinal fluid LGI1 antibody; c．Reasonable exclusion of other etiologies and other well-defined encephalitis syndromes (e.g., Bickerstaff brainstem encephalitis, acute disseminated encephalomyelitis, Hashimoto encephalopathy, primary CNS vasculitis, Rasmussen encephalitis);
4. Refractory AE: ineffective treatment with steroids and rituximab or other immunosuppressants, post-treatment mRS score≥2 (stable for at least 24 hours）;Recurrent AE: at least 2 months after 1st or 2nd line treatment, new symptoms or worsening of existing symptoms (mRS increase>1); 5）Doses of steroids and other immunosuppressants (e.g. azathioprine, mycophenolate mofetil, cyclophosphamide) should be stabilised for 4 weeks prior to enrolment; 6）Ability to obtain patient or proxy consent; 7）Women of childbearing potential should use effective contraception during treatment or avoid heterosexual intercourse for at least 3 months after the last dose of talitacicept;

Exclusion Criteria:

1. History of other autoimmunity such as SLE, RA, SS. Patients with hyperthyroidism and hypothyroidism cannot be excluded;
2. Abnormal laboratory indicators, including but not limited to the following indicators:

   White blood cell count<3×10^9 /L Neutrophil count<1.5×10^9 /L Hemoglobin<85g/L Blood platelet count<80×10^9 /L Serum creatinine>1.5×ULN TBil(total bilirubin) >1.5×ULN ALT>3× ULN AST>3× ULN Alkaline phosphatase>2× ULN Creatine kinase>5× ULN
3. Evidence of active infection such as shingles, HIV or active tuberculosis, etc.
4. Currently have active hepatitis or have severe liver disease and a history of it.

   * Patiens with abnormal Hepatitis B test as follows should be excluded: HbsAg positive; HbsAg negative but HbcAb positive, and HBV-DNA positive. Whereas patients with HbsAg negative but HbcAb positive, and HBV-DNA negative can be included.
   * Exclude patients who are positive for hepatitis C antibodies ;
5. Uncontrolled diabetes mellitus: Glycosylated hemoglobin>9.0% or fasting blood glucose≥11.1mmol/L;
6. Received any live vaccine within 3 months prior to enrollment or planned to receive any vaccine during the study;
7. Received rituximab or other biological therapies within 1 month prior to enrollment;
8. Malignancy;
9. Allergic to human biological products;
10. Participated in any clinical trial within 28 days prior to enrollment or within 5 times the half-life of the investigational drug participating in the clinical trial
11. Patients who plan to have children during the trial, or who are pregnant or breastfeeding;
12. Alcohol or drug abuse/addiction is known to have an impact on compliance with trial requirements;
13. Patients who are deemed unsuitable for the trial by the investigator (e.g., those with severe mental disorders).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
the change of mRS score | from baseline at week 24
  Refractory encephalitis: rate of patients with mRS score <2 or mRS score improvement of ≥2 points from baseline at week 24; Recurrent encephalitis: proportion of patients with no recurrence and [mRS score <2 or mRS score improvement of ≥2 points from baseline at week 24.
  mRS score vary from 0-6 score and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jiawei Wang, Study Director — Beijing Tong Ren Hospital
Locations (1):
- Beijing Tongren Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No